CLINICAL TRIAL: NCT04056247
Title: PROPHETIC - Predicting Responsiveness in Oncology Patients Based on Host Response Evaluation During Anti Cancer Treatments
Brief Title: Predicting Responsiveness in Oncology Patients Based on Host Response Evaluation During Anti Cancer Treatments
Acronym: PROPHETIC
Status: Active, not recruiting | Type: Observational
Sponsor: OncoHost Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: OH-HRPP-001
Record Dates: First submitted 2019-08-11; First posted 2019-08-14 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-07

CONDITIONS: Stage IV Non-small Cell Lung Cancer; Stage IV Malignant Melanoma; Stage IV Small Cell Lung Cancer; Stage III Unresectable Non-Small Cell Lung Cancer; Stage IIIb-d Malignant Melanoma
Keywords: Non-small Cell Lung Cancer; Small Cell Lung Cancer; Malignant Melanoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma; Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Stage IV NSCLC patients: Stage IV NSCLC patients treated with ICI or a combination of ICI and chemotherapy in any line of treatment, or with chemotherapy as a first line treatment.
  Interventions: Other: Plasma sample collection
- Stage III unresectable NSCLC patients: Patients with Stage III unresectable NSCLC treated with ICI therapy or ICI in combination with chemotherapy
  Interventions: Other: Plasma sample collection
- Stage IV malignant melanoma patients: Stage IV malignant melanoma patients treated with any regimen that includes ICI therapy as a monotherapy or in combination with targeted therapy in any line of treatment. In specific sites, Stage IV melanoma patients treated with targeted therapy (as a reference population).
  Interventions: Other: Plasma sample collection
- Stage IIIb-d malignant melanoma patients: Stage IIIb-d malignant melanoma patients treated with any regimen that includes ICI therapy as monotherapy or in combination with targeted therapy as adjuvant therapy.
  Interventions: Other: Plasma sample collection
- Stage IV SCLC patients: Stage IV SCLC patients treated with any regimen of ICI, chemotherapy or combination of ICI and chemotherapy in any line of treatment.
  Interventions: Other: Plasma sample collection

INTERVENTIONS:
Other: Plasma sample collection — Collect at least two plasma samples

SUMMARY:
The PROPHETIC study is a prospective, multi-center, international clinical study aimed at developing an algorithm to predict patient outcomes. The study involves analyzing the proteomic profiles of patients undergoing therapy to assess the likelihood of clinical benefit from their prescribed treatment. Blood samples are collected prior to and during the treatment period and analyzed as part of the ongoing development of thealgorithm.

DETAILED DESCRIPTION:
The goal of this research study is to develop an algorithm that predicts the patient's treatment outcome.This algorithm will serve as a tool for physicians when making treatment decisions, specifically for stage IV NSCLC and malignant melanoma patients receiving anti-cancer treatments. The investigators also aim to identify the metabolic pathways that could lead to better therapeutic options. The patients will be given their treatment according to the institute's standard of care. The patients will provide two blood samples and clinical data will be collected from their medical records.

In the first part of the trial, the data obtained from the blood samples and the medical records of the patients will be used to develop the prediction algorithm, and in the second part of the trial, the algorithm will be validated by comparing the objective response rate of the patients to the theoretical response prediction of the algorithm.

ELIGIBILITY:
Inclusion criteria

* Provision of informed consent prior to any study-specific procedures.
* Male or female aged at least 18 years.
* ECOG PS - 0/1-2
* Normal hematologic, renal and liver function:

  1. Absolute neutrophil count higher than 1500/mm3
  2. Platelets count higher than 100,000/mm3
  3. haemoglobin higher than 9 g/dL
  4. Creatinine concentration ≤1.4 mg/dL, or creatinine clearance higher than 40 mL/min
  5. Total bilirubin lower than 1.5 mg/dL, ALT and AST levels ≤ 3 times above the upper normal limit.
* At least one measurable lesion in order to enable the assessment of the response (except for stage IIIb-d malignant melanoma patients).

Exclusion Criteria:

* Concurrent and/or other active malignancy that has required systemic treatment within 2 years of first dose of study drug
* Generalized impairment or mental incompetence that would render the patient unable to understand his/her participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Stage IV NSCLC patients treated with ICI or a combination of ICI and chemotherapy in any line of treatment, or with chemotherapy as a first line treatment.
  2. Stage III unresectable NSCLC patients treated with ICI therapy or ICI in combination with chemotherapy.
  3. Stage IV malignant melanoma patients treated with any regimen that includes ICI therapy as a monotherapy or in combination with targeted therapy in any line of treatment. In specific sites, Stage IV melanoma patients treated with targeted therapy (as a reference population).
  4. Stage IIIb-d malignant melanoma patients treated with any regimen that includes ICI therapy as monotherapy or in combination with targeted therapy as adjuvant therapy.
  5. Stage IV SCLC patients treated with any regimen of ICI, chemotherapy or combination of ICI and chemotherapy in any line of treatment.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2029-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Measured biological features at baseline (pre-treatment) and after 1st dose administration (on-treatment) and during treatment (optional) | Measured biological features are analyzed in samples taken at baseline (prior treatment) and after the 1st dose administration (on-treatment) and during treatment (optional)
  Biological features are analyzed in biological samples taken from the patients as part of the study
Overall response as determined by RECIST 1.1 or any other validated clinical scales for response, every 3 months or according to the standard of care | Every 3 months or according to the standard of care
  Overall response as determined by RECIST 1.1 or any other validated clinical scales for response, every 3 months or according to the standard of care
Progression Free Survival (PFS) | At progression during treatment
  Collect Progression Free Survival (PFS) dates
Overall survival or last follow-up | Overall survival or last follow-up
  Collect overall survival or last follow-up dates

SECONDARY OUTCOMES:
Adverse Events (AE) | Adverse events (AE) during treatment and until the end of study
  AE to treatment, as reported by the patient

CONTACTS AND LOCATIONS:
Overall Officials: Alona Zer, MD, Principal Investigator — Rambam Health Care Campus; Michal Lotem, MD, Principal Investigator — Hadassah Medical Organization; Jair Bar, MD, Principal Investigator — Sheba Medical Center; Maya Gottfried, MD, Principal Investigator — Meir Medical Center; Abed Agbaria, MD, Principal Investigator — Bnai Zion Medical Center; Ido Wolf, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center; Mahmud Abu-Amana, MD, Principal Investigator — haemek medical center; Rivka Katsenelson, MD, Principal Investigator — Kaplan Medical Center; Alexander Yakobson, MD, Principal Investigator — Soroka University Medical Center; Tatiana Harkovsky, MD, Principal Investigator — Barzilai Medical Center; Mor Moskovitz, MD, Principal Investigator — Rabin Medical Center; Elizabeta Dudnik, MD, Principal Investigator — Assuta Medical Center; Raya Leibowitz, MD, Principal Investigator — Assaf-Harofeh Medical Center; Adam Berger, MD, Principal Investigator — Rutgers Cancer Institute; Jose Lutzky, MD, Principal Investigator — University of Miami; Antony Magliocco, MD, Principal Investigator — Protean BioDiagnostics; Gillian Price, MD, Principal Investigator — Aberdeen Royal Infirmary; Helen Cheley, Principal Investigator — Swansea Bay UHB - Cancer Institute; Louise Medley, MD, Principal Investigator — Torbay and South Devon NHS foundation; Tom Geldart, MD, Principal Investigator — Royal Bournemouth General Hospital Dorset; Anirban Chatterjee, MD, Principal Investigator — The Shrewsbury and Telford Hospital; Sean Brown, MD, Principal Investigator — Gloucestershire Hospitals NHS Foundation Trust; Andreas Polychronis, MD, Principal Investigator — Mount Vernon Cancer Centre; Andreas Polychronis, MD, Principal Investigator — Lister Hospital; Ari VanderWalde, MD, Principal Investigator — West Clinic; Davika Das, MD, Principal Investigator — VAHCS Birmingham; Alison Brewster, MD, Principal Investigator — Withybush Hospital Hawl Dda University Health Board; Adam Hassani, Principal Investigator — Sunderland Royal Hospital; Adam Hassani, MD, Principal Investigator — South Tyneside District; Andrew Conn, MD, Principal Investigator — Bradford Teaching Hospitals; Yanyan Lou, MD, Principal Investigator — Mayo Clinic; Igor Puzanov, MD, Principal Investigator — Roswell Park; Ernesto Bustinza, MD, Principal Investigator — Florida Cancer Specialists and Research Institute; Huang Quillan, MD, Principal Investigator — Michael E. DeBakey VA Medical Center; Ronnie Shapira Frommer, MD, Principal Investigator — Sheba Medical Center; Astrid Ammendola, MD, Principal Investigator — Asklepios Klinik Gauting GmbH; Petros Christopoulos, MD, Principal Investigator — Thoraxklinik-Heidelberg gGmbH; Marina Messinger, MD, Principal Investigator — Northwest Community Healthcare; Sunil Patel, MD, Principal Investigator — CHRISTUS St. Michael Health System; Bharat P Jenigiri, MD, Principal Investigator — Physicians Clinic of Iowa; David Vecente, MD, Principal Investigator — Hospital Universitario Virgen Macarena; Eugenie Younger, MD, Principal Investigator — Gloucestershire Hospitals NHS Foundation Trust
Locations (41):
- United States (12):
  - Birmingham VAHCS, Birmingham, Alabama
  - Mayo Clinic, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Florida Cancer Specialist and Research Institute, Orlando, Florida
  - Protean Biodiagnosics, Orlando, Florida
  - Northwest Community Healthcare, Rolling Meadows, Illinois
  - Helen Nassif Community Cancer Center, Cedar Rapids, Iowa
  - Rutgers Cancer Institute, New Brunswick, New Jersey
  - Roswell Park, Buffalo, New York
  - West Clinic, Germantown, Tennessee
  - Michael E. Debakey VA Medical Center, Houston, Texas
  - 151-Christus Health St. Michael, Texarkana, Texas
- Germany (2):
  - Asklepois, Gauting
  - Thoraxklinik Heidelberg gGmbH, Heidelberg
- Israel (14):
  - Haemek Medical Center, Afula
  - Barzilai Medical Center, Ashkelon
  - Soroka Medical Center, Beersheba
  - Shamir Medical Center, Be’er Ya‘aqov
  - Bnai Zion Medical Center, Haifa
  - Rambam Medical Center, Haifa
  - Hadassah Medcial Center, Jerusalem
  - Meir medical center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Assuta Medical Cetner, Tel Aviv
  - Sheba Medical Center, Tel Aviv
  - Sourasky Medical Center, Tel Aviv
  - Sheba medical center, Tel Litwinsky
- 044 Hospital Universitario Virgen Macarena, Seville, Spain
- United Kingdom (12):
  - Aberdeen Royal Infirmary, Aberdeen
  - Royal Bournemouth General Hospital, Bournemouth
  - Bradford Teaching Hospitals, Bradford
  - Cheltenham General Hospital, Cheltenham
  - Withybush Hospital, Haverfordwest
  - Mount Vernon Cancer Centre, Northwood
  - The Shrewsbury and Telford Hospital, Shrewsbury
  - South Tyneside, South Shields
  - Lister Hospital, Stevenage
  - Sunderland Royal Hospital, Sunderland
  - Swansea Bay UHB Singleton Hospital, Swansea
  - Torbay Hospital, Torquay

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shaked Y. Balancing efficacy of and host immune responses to cancer therapy: the yin and yang effects. Nat Rev Clin Oncol. 2016 Oct;13(10):611-26. doi: 10.1038/nrclinonc.2016.57. Epub 2016 Apr 26. PMID 27118493
- [Background] Shaked Y, Kerbel RS. Antiangiogenic strategies on defense: on the possibility of blocking rebounds by the tumor vasculature after chemotherapy. Cancer Res. 2007 Aug 1;67(15):7055-8. doi: 10.1158/0008-5472.CAN-07-0905. PMID 17671170
- [Background] Shaked Y, Bocci G, Munoz R, Man S, Ebos JM, Hicklin DJ, Bertolini F, D'Amato R, Kerbel RS. Cellular and molecular surrogate markers to monitor targeted and non-targeted antiangiogenic drug activity and determine optimal biologic dose. Curr Cancer Drug Targets. 2005 Nov;5(7):551-9. doi: 10.2174/156800905774574020. PMID 16305351
- [Derived] Christopoulos P, Harel M, McGregor K, Brody Y, Puzanov I, Bar J, Elon Y, Sela I, Yellin B, Lahav C, Raveh S, Reiner-Benaim A, Reinmuth N, Nechushtan H, Farrugia D, Bustinza-Linares E, Lou Y, Leibowitz R, Kamer I, Zer Kuch A, Moskovitz M, Levy-Barda A, Koch I, Lotem M, Katzenelson R, Agbarya A, Price G, Cheley H, Abu-Amna M, Geldart T, Gottfried M, Tepper E, Polychronis A, Wolf I, Dicker AP, Carbone DP, Gandara DR. Plasma Proteome-Based Test for First-Line Treatment Selection in Metastatic Non-Small Cell Lung Cancer. JCO Precis Oncol. 2024 Mar;8:e2300555. doi: 10.1200/PO.23.00555. PMID 38513170